CLINICAL TRIAL: NCT02557633
Title: A Pre-season, Single Site, Single-blind, Parallel Group, Randomized Study to Determine the Tolerability and Safety of Two New Cumulative Doses of Modified Grass Allergens Adsorbed to L-tyrosine With Monophosphoryl Lipid A Adjuvant (Corixa), Phenol Preserved (Grass MATA MPL); Allergy Therapeutics, (UK) Ltd., Compared With Placebo in Patients With Seasonal Allergic Rhinoconjunctivitis Due to Grass Pollen Allergy.
Brief Title: A Study of Tolerability and Safety of Two New Doses of Grass MATA MPL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Collaborators: Inflamax Research Incorporated (Industry); Metronomia Clinical Research GMBH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrassMATAMPL102
Record Dates: First submitted 2015-09-15; First posted 2015-09-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): 2% w/v L-Tyrosine
  Interventions: Biological: Placebo
- Grass MATA MPL 10200 SU (Experimental): Grass MATA MPL cumulative dose 10200 SU given as six injections of placebo, placebo, 600SU, 1600SU, 4000SU and 4000SU.
  Interventions: Biological: Grass MATA MPL 10200
- Grass MATA MPL 18200 SU (Experimental): Grass MATA MPL cumulative dose 18200 SU given as six injections of 600SU, 1600SU, 4000SU, 4000SU, 4000SU and 4000SU.
  Interventions: Biological: Grass MATA MPL 18200

INTERVENTIONS:
Biological: Grass MATA MPL 10200
  Arms: Grass MATA MPL 10200 SU
Biological: Grass MATA MPL 18200
  Arms: Grass MATA MPL 18200 SU
Biological: Placebo
  Arms: Placebo

SUMMARY:
There is increasing evidence that the effectiveness of allergy immunotherapy to control symptoms of rhinoconjunctivitis is related to the cumulative dose of allergen or allergoid administered during a single regimen of subcutaneous (SC) injections or of sublingual administration.

Two new cumulative doses of the Grass MATA MPL 10200 and 18200 SU (Standardized Units) are being developed to compare with the current dose of 5100 SU. The purpose of this study is to evaluate the tolerability and safety of these two new cumulative dose regimens of Grass MATA MPL compared with placebo in patients with seasonal allergic rhinoconjunctivitis (SAR) due to grass pollen, to enable selection of the best dose to go into a larger scale study to assess the efficacy and safety of the higher cumulative doses.

DETAILED DESCRIPTION:
Structure: Single center, parallel group, single-blind, randomized study There will be three treatment groups, two groups receiving a different, cumulative dose of Grass MATA MPL and the third group receiving placebo only.

Duration: The duration of the study from screening to final visit after treatment is expected to be approximately 7 weeks. There will be a telephone follow up at 1, 3, 6 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a positive skin prick test for grass pollen allergen.
* Positive skin prick test to positive histamine control
* Negative skin prick test to negative control
* Specific IgE for grass pollen as documented by radioallergosorbent or equivalent test with class ≥ 2
* History of at least 2 seasons of moderate to severe seasonal rhinoconjunctivitis due to an IgE - mediated allergy to pollen from grass
* Males or non-pregnant, non-lactating females who are:

  * Post-menopausal (defined as at least 12 months natural spontaneous amenorrhea or at least 6 weeks following surgical menopause, i.e. bilateral oophorectomy)
  * Naturally or surgically sterile (hysterectomy; bilateral oophorectomy; bilateral tubal ligation with surgery at least 6 weeks prior to study initiation)
  * Of childbearing potential - with negative urinary and serological pregnancy test and use at least one of the following contraception methods:
  * Stable hormonal contraceptive for ≥ 90 days prior to Visit 1 and at least 7 days after the final injection. If < 90 days prior to the study, additional use of a double barrier method until 90 days reached is required.
  * Placement of an intrauterine device (IUD) or intrauterine system
  * Use of barrier methods of contraception (e.g., condom or occlusive cap) with spermicidal foam/gel/film/cream /suppository
  * Use of double barrier methods of contraception (e.g., male condom with diaphragm, male condom with cervical cap)
* Patients who are normally active and otherwise judged to be in good health
* Patients must be willing and able to attend required study visits.
* Patients must be able to follow instructions.
* Patients must be willing and able to give written informed consent and must provide this consent.

Exclusion Criteria:

* Symptoms outside the grass pollen season due to a perennial and/or non-grass seasonal allergen, if the patient is unable to avoid the offending allergen.
* Concurrent disease that might complicate or interfere with investigation or evaluation of the study medications or the skin prick test result, such as:

  * Any ocular disorder (other than allergic conjunctivitis) including presumed infectious ocular disease (bacterial, fungal, viral, etc.), which could interfere with the evaluation of the study medication Rhinitis medicamentosa
  * Documented evidence of acute or significant chronic sinusitis, upper or lower respiratory tract infection within 30 days before Visit 2 as determined by the Investigator
  * Asthma, with the exception of mild intermittent asthma
  * Emergency room visit or admission for asthma in the 12 months prior to Visit 1 or history of a life-threatening asthma attack ever
  * Presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence
  * Presence of emphysema or bronchiectasis
* Auto-immune disease, cancer, or concomitant illness that in the opinion of the Investigator would pose a safety risk or compromise the interpretation of study results
* Use of oral, intramuscular, intravenous corticosteroids, or potent or super-potent topical corticosteroids, from 30 days prior to screening up to Visit 8
* Presence of tattoos or other skin abnormalities in the upper arms which would prevent an accurate assessment of local skin reaction
* Allergy, hypersensitivity or intolerance to the excipients of the study medication
* Anaphylactic reactions to foods, insect venom, exercise, drugs or idiopathic anaphylaxis
* Immunodeficiency, including those who are on immunosuppressant therapy
* Recurrent idiopathic angioedema
* Tyrosine metabolism disorders, especially tyrosinemia and alkaptonuria
* β-blocker (including eye drops), monoamine oxidase medication
* Unable to receive epinephrine therapy (i.e., use of epinephrine is contraindicated)
* Clinical history of drug or alcohol abuse, at the Investigator's discretion, that would interfere with the patient's participation in the study
* Any clinically significant abnormal laboratory value (as determined by the Investigator) at Visit 1
* Study site staff or immediate relatives of study site staff or other individuals who would have access to the clinical study protocol or people considered as vulnerable or institutionalized
* Have undergone specific immunotherapy with comparable allergen extracts. An exception will be allowed if prior immunotherapy with comparable allergen was successful, symptoms reappeared some-time after stopping the immunotherapy, and the immunotherapy was completed ≥ 3 years before Visit 1
* Treatment with a preparation containing MPL® within 6 months prior to Visit 1.
* Participation in a clinical research study with an investigational medicinal product within 4 weeks of Visit 1 or concomitantly with this study, including the safety follow-up period up to 12 months following the last injection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of AEs | 8 weeks
  Aggregate of the number of AEs, adverse reaction complexes (ARCs; the total of treatment related injection site and systemic AEs experienced by a patient within a 24-hour period after an injection)
Premature discontinuation | 8 weeks
  The frequency of premature discontinuation from treatment or study due to AEs between the treatment groups

SECONDARY OUTCOMES:
AEs of special interest | one year
  The number and frequency of neuro-inflammatory or new onset autoimmune disease.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Higenbottam, DSc MD FRCP FFPM, Study Director — Allergy Therapeutics
Locations (2):
- United States (2):
  - Inflamax Research, Inc., Neptune City, New Jersey
  - Inflamx Research, Newark, New Jersey